CLINICAL TRIAL: NCT00083499
Title: Mutations in Genes Associated With Pentalogy of Cantrell
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040202; 04-H-0202
Record Dates: First submitted 2004-05-25; First posted 2004-05-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pentalogy of Cantrell
Keywords: Nonmuscle myosin IIB; Nonmuscle myosin IIA; Pentology of Cantrell; thoracoabdominal syndrdome; Nonmuscle Myosin IIC; Pentalogy of Cantrell; Non-muscle Myosin Heavy Chain Genes
MeSH Terms: conditions — Pentalogy of Cantrell; MYH9-Related Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Index cases
- Group 2: Relatives of Index Cases
- Group 3: Fetal tissue

SUMMARY:
This study will collect blood, urine, and other tissue samples from patients with Pentalogy of Cantrell (POC) and other inherited diseases that may involve mutations in non-muscle myosin II-B heavy chain (MYH10). We will also collect samples from the relatives of affected individuals. POC is a very rare disorder in which patients have a combination of severe defects of the middle of the chest including the sternum (breastbone), diaphragm, heart, and abdominal wall. The defect are apparent before birth or at birth.

Participants may undergo a medical evaluation that could include a medical history routine blood tests, urine collection, chest x-ray, and electrocardiogram. In addition, blood, urine, saliva, buccal swab or tissue samples may be collected for protein and gene studies. The blood is drawn through a very small needle placed in an arm vein. Children may choose to have a buccal (cheek) sample taken instead of blood draw. Buccal samples can be collected by a cheek swab, in which a soft brush is rubbed on the inside lining of the mouth, or by having the child hold a tablespoon of mouthwash in his or her mouth for a full minute and then spit the mouthwash into a container. In addition, tissue samples may be collected from patients if they undergoing any surgical procedures that may be required as part of their general medical care.

Some of the cells obtained from patients or their relatives may be used to establish cell lines (a living tissue sample) that can be grown in the laboratory and used for experiments.

...

DETAILED DESCRIPTION:
The purpose of this multisite protocol is to collect protein, DNA, and RNA from blood, sputum, urine and/or tissue samples from patients with the diagnosis of Pentalogy of Cantrell (POC) or other related syndromes in order to identify possible causative genes. We will use whole exome/genome sequencing of probands, their parents, and, if available, the affected relatives of probands to look for any exomic/genomic mutations that could be associated with this syndrome. We have produced a mouse model with the mutant mice exhibiting problems with ventral wall closure including extrathoracic location of the heart (ectopia cordis), and defects in the abdominal wall with protrusion of the guts and liver. The mice, which have a single amino acid substitution in nonmuslce myosin II-B, have severe defects in both the heart and brain, and resemble humans born with POC, who manifest these same abnormalities.

ELIGIBILITY:
* INCLUSION CRITERIA:

  i. Index Cases
  1. Those patients who have a diagnosis of POC or other related syndromes (as defined under Study Design) confirmed by telephone discussion between the investigators and the patient s physician.
  2. Outside Institutions- All ages will be included
  3. At the Clinical Center - Those subjects that are greater than or equal to 2 years of age and older.

ii. Relatives of Index Cases

1. We may obtain samples from family members and/or relatives of those individuals who have a diagnosis of POC or other related syndrome confirmed by telephone discussion between the investigators and the referring physician with knowledge of the index case.
2. Outside Institutions - All ages will be included. At the Clinical Center - Those subjects that are greater than or equal to 2 years of age and older

iii. Fetal tissue:

1. We may obtain samples from patients with a fetal diagnosis of POC or other related syndrome with diagnosis confirmed by telephone discussion between the investigators and the referring physician.
2. Research use of the fetal tissue in accordance to NIH Division of Intramural Research (DIR) Program fetal tissue policy guidelines:

   1. No profits will be involved;
   2. NIH researchers will have no involvement in the termination of pregnancy, and
   3. The tissue must be obtained in accordance with Federal, state, and local law including those that govern basic research using human fetal tissue and research involving the transplantation of fetal tissue.

EXCLUSION CRITERIA:

Subjects seen at the Clinical Center - Those subjects that are less than or equal to 2 years of age and older.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2004-09-15 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Identify the gene(s) mutation (s) that causes Pentalogy of Cantrell | ongoing
  Identification of novel genes related to Pentalogy of Cantrell

SECONDARY OUTCOMES:
Since mutations in NM IIB may not be the sole cause of POC, we also intend to identify any other gene(s) mutation(s) that might be thecause of POC. | Ongoing
  Identifying any other gene(s) mutation(s) that might be the cause of POC.
We may wish to procure tissues from patients with nonmuscle myosin IIA and IIC mutations in order to study the mechanism underlyingthese abnormalities. | Ongoing
  Studying the mechanism underlying these abnormalities in procuredtissues from patients with nonmuscle myosin IIA and IIC mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Adelstein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Ma X, Adelstein RS. In vivo studies on nonmuscle myosin II expression and function in heart development. Front Biosci (Landmark Ed). 2012 Jan 1;17(2):545-55. doi: 10.2741/3942. PMID 22201759
- [Background] Ma X, Adelstein RS. The role of vertebrate nonmuscle Myosin II in development and human disease. Bioarchitecture. 2014;4(3):88-102. doi: 10.4161/bioa.29766. Epub 2014 Aug 6. PMID 25098841
- [Background] Ma X, Adelstein RS. A point mutation in Myh10 causes major defects in heart development and body wall closure. Circ Cardiovasc Genet. 2014 Jun;7(3):257-65. doi: 10.1161/CIRCGENETICS.113.000455. Epub 2014 May 13. PMID 24825879
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-H-0202.html